CLINICAL TRIAL: NCT03081156
Title: An Investigator Initiated, Randomized, Double Blind, Placebo Controlled Study to Assess the Effect of Glycopyrrolate/Formoterol on Exercise Tolerance and Dynamic Hyperinflation in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: The Effect of BEVESPI AEROSPHERE ® Therapy on Exercise Tolerance in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: William Stringer, md (Other)
Responsible Party: Sponsor-Investigator, William Stringer, md, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21752-01
Record Dates: First submitted 2017-03-09; First posted 2017-03-16 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: chronic obstructive pulmonary disease (COPD); exercise intolerance; dynamic hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Cross-Over Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glycopyrrolate/Formoterol Inhaler then Placebo Inhaler (Active Comparator): Participants receive the Glycopyrrolate/Formoterol inhaler for a two week period. After a two week washout, the participants then received a placebo Glycopyrrolate/Formeterol inhaler for two weeks.
  Interventions: Drug: Glycopyrrolate / Formoterol Inhaler vs Placebo Inhaler
- Placebo Inhaler then Glycopyrrolate/Formeterol Inhaler (Placebo Comparator): Treatment for 2 weeks with a placebo Glycopyrrolate/Formoterol inhaler. After a two week washout, the participant then received two weeks of the Glycopyrrolate/Formoterol inhaler.
  Interventions: Drug: Glycopyrrolate / Formoterol Inhaler vs Placebo Inhaler

INTERVENTIONS:
Drug: Glycopyrrolate / Formoterol Inhaler vs Placebo Inhaler — Exercise Tolerance
  Other Names: Bevespi AEROSPHERE

SUMMARY:
The objective of the study is to determine if a dual inhaled bronchodilator (Glycopyrrolate/Formoterol) is effective in increasing exercise time relative to placebo in patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Enrolled patients with COPD will be randomized to receive either a dual bronchodilator (Glycopyrrolate/Formoterol) or placebo inhaler, and then crossed over to receive the opposite intervention. The study will consist of two treatment periods of two weeks, seperated by a washout period of two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a clinical diagnosis of chronic obstructive pulmonary disease (COPD) and must meet the following criteria:

   1. Stable state of their disease with no exacerbation (antibiotics, oral steroids, ER visit, or hospitalization for COPD) within the previous 4 weeks; and
   2. At visit 1 Spirometric Values must demonstrate a post-bronchodilator FEV1 between 35% and 80% of predicted normal and a post-bronchodilator FEV1/FVC <70%. [The rationale for the lower limit is to exclude patients unlikely to tolerate withholding of long acting bronchodilators. The rationale for the upper limit is to exclude patients unlikely to be limited in their exercise tolerance by hyperinflation and air trapping.]
2. Male or female patients, between 40 and 80 years (inclusive) of age.
3. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years.
4. Patients must be able to perform technically acceptable pulmonary function tests and a symptom-limited cardiopulmonary cycle ergometry test.
5. Patients must be able to inhale medication in an acceptable manner from the metered dose inhalers used in this study.

Exclusion Criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study.
2. Patients with a documented personal history of childhood asthma, a clinical presentation consistent with asthma, and a family history of asthma. For patients with allergic rhinitis, atopy, or prior allergy treatment, medical records will be obtained to verify that the patient does not have asthma. The final determination on the possibility of an overlap condition [Asthma-COPD Overlap Syndrome, (Postma and Rabe, 2015)], and thus, appropriateness for entry into the study, will be the principal investigator's decision.
3. Patients with any of the following conditions:

   1. A history of myocardial infarction within 1 year of screening visit.
   2. Unstable or life-threatening cardiac arrhythmia.
   3. Hospitalized for heart failure within the past year.
   4. Known active tuberculosis.
   5. A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within the past 6 months (patients with treated local skin tumors are allowed).
   6. A history of life-threatening COPD exacerbation requiring intubation.
   7. A history of cystic fibrosis.
   8. Clinically significant and active bronchiectasis.
   9. A history of alcohol or drug abuse within the past year.
   10. Any contraindications for exercise testing as outlined below (see contraindications to exercise).
   11. Patients who have undergone thoracotomy with pulmonary resection in the past year.
4. Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
5. Patients who regularly use daytime oxygen therapy for more than 6 hours per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits and exercise testing.
6. Patients who desaturate to SpO2 <80% on screening incremental exercise testing.
7. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
8. Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea, such as arthritis in the leg, angina pectoris or claudication or morbid obesity.
9. Patients with a constant power cycle ergometry endurance time less than 4 or greater than 8 minutes after work rate adjustment procedures (described below).
10. Patients who have taken an investigational drug within one month or six half-lives (whichever is greater) prior to screening visit (Visit 1).
11. Pregnant or nursing women.
12. Women of childbearing potential who are not using a highly effective method of birth control. Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
13. Patients who are currently participating in another interventional study.
14. Patients who are unable to comply with pulmonary medication restrictions (washout of any LABA/LAMA) prior to randomization.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stringer, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stringer WW, Porszasz J, Cao M, Rossiter HB, Siddiqui S, Rennard S, Casaburi R. The effect of long-acting dual bronchodilator therapy on exercise tolerance, dynamic hyperinflation, and dead space during constant work rate exercise in COPD. J Appl Physiol (1985). 2021 Jun 1;130(6):2009-2018. doi: 10.1152/japplphysiol.00774.2020. Epub 2021 Apr 29. PMID 33914661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty participants were screened for eligibility.
Pre-assignment Details: 52 of the 60 participants signed informed consent., however, only 48 were randomized. 4 participants withdrew consent in the pre-randomization period.
Groups:
- Glycopyrrolate/Formoterol Inhaler First, Then Placebo: First Intervention: Bevespi Aerosphere (Glycopyrrolate/Formoterol) twice daily for 14 days, then washout for 14 days, then Second Intervention: Placebo Inhaler twice daily for 14 days.
- Placebo First, Then Glycopyrrolate/Formoterol Inhaler: First Intervention: Placebo Inhaler twice daily for 14 days, then washout for 14 days, then Second Intervention: .Bevespi Aerosphere (glycopyrrolate/Formoterol) twice daily for 14 days
Period: Overall Study
Arm/Group | Glycopyrrolate/Formoterol Inhaler First, Then Placebo | Placebo First, Then Glycopyrrolate/Formoterol Inhaler
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Male or Female patients between 40 and 80 years old with a clinical diagnosis of COPD (post bronchodilator FEV1 to FEV ratio <0.7).
Groups:
- Participants Received Glycopyrrolate/Formoterol Inhaler Then Placebo Inhaler: Participants received 14 days of the the Glycopyrrolate/Formoterol Inhaler. They They then washed out for 14 days, then received a placebo Inhaler for 14 days.
  At the end of the first and second 14 day intervention period, the participants performed a constant work rate bicycle ergometer exercise test to determine the effect on exercise tolerance.
  The outcome is time in seconds compared to their baseline value.
- Participants Received Placebo Inhaler Then Glycopyrrolate/Formoterol Inhaler: Participants received 14 days of the a placebo inhaler. They then washed out for 14 days, then received 14 days of a Glycopyrrolate/Formoterol Inhaler
- Total: Total of all reporting groups
Arm/Group | Participants Received Glycopyrrolate/Formoterol Inhaler Then Placebo Inhaler | Participants Received Placebo Inhaler Then Glycopyrrolate/Formoterol Inhaler | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.7) | 62.3 (8.1) | 62.9 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Time (Seconds) During Cycle Ergometer Exercise.
Description: To determine the magnitude of exercise time improvement (seconds) with BEVESPI AEROSPHERE ® (Glycopyrrolate/Formeterol) relative to placebo during high intensity, constant work rate cycle ergometer exercise in COPD patients.
Time Frame: 8-12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Glycopyrrolate/Formoterol Inhaler: Treatment for 2 weeks with Bevespi Aerosphere (Glycopyrrolate/Formoterol) inhaler to determine the effect on exercise tolerance using a constant work rate bicycle ergometer exercise test. The outcome is time in seconds compared to their baseline value.
  Glycopyrrolate / Formoterol: Exercise Tolerance
- Placebo: Treatment for 2 weeks with a placebo Bevespi Aerosphere (Glycopyrrolate/Formoterol) inhaler to determine the effect on exercise tolerance using a constant work rate bicycle ergometer exercise test. The outcome is time in seconds compared to their baseline value.
  Glycopyrrolate / Formoterol: Exercise Tolerance
Arm/Group | Glycopyrrolate/Formoterol Inhaler | Placebo
Number analyzed (Participants) | 48 | 48
seconds | 382.50 (184.17) | 328 (115.45)

2. Secondary Outcome: VD/VT as Determined by Transcutaneous CO2 Measurement (tcpCO2) During Constant Work Rate Cycle Ergometer Exercise.
Description: To determine if the VD/VT can be reliably assessed during constant work rate exercise using transcutaneous CO2 measurement (tcpCO2) and, if so, if BEVESPI AEROSPHERE ® (Glycopyrrolate/Formeterol) results in a reduction in VD/VT relative to placebo at isotime during high intensity constant work rate exercise in COPD patients.
Time Frame: 8 to 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Glycopyrrolate/Formoterol Inhaler | Placebo
Number analyzed (Participants) | 48 | 48
ratio | 0.28 (.01) | .028 (.01)

ADVERSE EVENTS:
Time Frame: 8 to 12 weeks
Description: Same Definition.
Arm/Group | Glycopyrrolate/Formoterol Inhaler | Placebo
All-Cause Mortality (participants affected / at risk) | 48/48 | 48/48
Serious Adverse Events (participants affected / at risk) | 6/48 | 3/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrrolate/Formoterol Inhaler (N=48) | Placebo (N=48)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) — Dyspnea with Exercise Testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT03081156/Prot_SAP_003.pdf
  • Informed Consent Form (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT03081156/ICF_004.pdf